CLINICAL TRIAL: NCT02399085
Title: A Phase II, Single-Arm, Open-Label, Multicentre Study to Evaluate the Safety and Efficacy of Lenalidomide Combined With MOR00208 in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R-R DLBCL)
Brief Title: Open Label Study to Evaluate the Safety and Efficacy of Lenalidomide With MOR00208 in Patients With R-R DLBCL
Acronym: L-MIND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR208C203; 2014-004688-19 (EudraCT Number)
Record Dates: First submitted 2015-03-13; First posted 2015-03-26 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; Efficacy; MOR00208; Tafasitamab; lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Tafasitamab (MOR00208) + lenalidomide (LEN) (Experimental): MOR00208:
  MOR00208 was administered via IV infusion at a dose of 12 mg/kg. For the first three cycles (Cycles 1 to 3) of the study each cycle consisted of a MOR00208 infusion on Day 1, Day 8, Day 15 and Day 22 of the cycle.
  Additionally, a loading dose was administered on Day 4 of Cycle 1. Thereafter MOR00208 was administered on a bi-weekly (every 14 days) basis with infusions on Day 1 and Day 15 of each 28-day cycle.
  LEN:
  Participants self-administered a starting dose of 25 mg oral LEN daily on Days 1-21 of each cycle, for up to 12 cycles in total. LEN dose could be modified in a de-escalating fashion or discontinued based upon clinical and laboratory findings.
  On days when both study drugs were given together, LEN was administered prior to MOR00208.
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Tafasitamab — 12 mg/kg
  Other Names: MOR00208
Drug: Lenalidomide — 25 mg
  Other Names: LEN; Revlimid®

SUMMARY:
This is a Phase II, Single-Arm, Open-Label, Multicentre Study to Evaluate the Safety and Efficacy of Lenalidomide Combined with MOR00208 in Participants with Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R-R DLBCL).

DETAILED DESCRIPTION:
The aim of this single-arm, multicentre, open-label Phase II study is to evaluate the Lenalidomide (LEN) combined with Tafasitamab (MOR00208) in adult participants with DLBCL who had relapsed after or were refractory to at least one, but no more than three previous systemic regimens administered for the treatment of their DLBCL and who were not candidates for high-dose chemotherapy and subsequent Autologous stem cell transplants and were thus considered to have exhausted their therapeutic options. One prior therapy line had to include an anti-CD20 targeted therapy (e.g., rituximab [RTX]).

MOR00208 and LEN were administered for up to 12 cycles (28 days each), followed by MOR00208 monotherapy until progression, in participants with at least stable disease or a better response.

ELIGIBILITY:
Major Inclusion Criteria:

1. Age >18 years
2. Histologically confirmed diagnosis of DLBCL
3. Tumour tissue for central pathology review and correlative studies had to be provided.
4. Participants must had:

   * relapsed and/or refractory disease
   * at least one bidimensionally measurable, PET positive disease site (transverse diameter of ≥1.5 cm and perpendicular diameter of ≥1.0 cm at baseline)
   * received at least one, but no more than three previous systemic regimens for the treatment of DLBCL and one therapy line must had included a CD20-targeted therapy
   * Eastern Cooperative Oncology Group 0 to 2
5. Participants were not considered in the opinion of the investigator eligible, or participants unwilling to undergo intensive salvage therapy including ASCT
6. Participants had to meet the following laboratory criteria at screening:

   * absolute neutrophil count ≥1.5 × 10˄9/L
   * platelet count ≥90 × 10˄9/L
   * total serum bilirubin ≤2.5 × ULN or ≤5 × ULN in cases of Glibert's Syndrome or liver involvement by lymphoma
   * alanine transaminase, aspartate aminotransferase and alkaline phosphatase ≤3 × ULN or <5 × ULN in cases of liver involvement
   * serum creatinine clearance ≥60 mL/minute
7. Females of childbearing potential (FCBP) must:

   * not be pregnant
   * refrain from breastfeeding and donating blood or oocytes
   * agreed to ongoing pregnancy testing
   * committed to continued abstinence from heterosexual intercourse, or agree to use and be able to comply with the use of double-barrier contraception
8. Males (if sexually active with a FCBP) had to

   * use an effective barrier method of contraception
   * refrain from donating blood or sperm
9. In the opinion of the investigator the participants had to:

   * be able and willing to receive adequate prophylaxis and/or therapy for thromboembolic events
   * be able to understand, give written informed consent and comply with all study-related procedures, medication use, and evaluations
   * had no history of noncompliance in relation to medical regimens or not be considered potentially unreliable and/or uncooperative
   * be able to understand the reason for complying with the special conditions of the pregnancy prevention risk management plan and gave written acknowledgement of this.

Major Exclusion Criteria:

1. Participants who had:

   * other histological type of lymphoma
   * primary refractory DLBCL
   * a history of "double/triple hit" genetics
2. Participants who had, within 14 days prior to Day 1 dosing:

   * not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy or other lymphoma specific therapy
   * underwent major surgery or suffered from significant traumatic injury
   * received live vaccines.
   * required parenteral antimicrobial therapy for active, intercurrent infections
3. Participants who:

   * had, in the opinion of the investigator, not recovered sufficiently from the adverse toxic effects of prior therapies
   * were previously treated with CD19-targeted therapy or immunomodulatory drugs (IMiDs)® (e.g., thalidomide, LEN)
   * had a history of hypersensitivity to compounds of similar biological or chemical composition to MOR00208, IMiDs® and/or the excipients contained in the study drug formulations
   * had undergone ASCT within the period ≤ 3 months prior to the signing of the Informed Consent Form. Patients who had a more distant history of ASCT had to exhibit full haematological recovery before enrolment into the study
   * had undergone previous allogenic stem cell transplantation
   * had a history of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia or were at a high risk for a thromboembolic event in the opinion of the investigator and who were not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period
   * concurrently used other anti-cancer or experimental treatments
4. Prior history of malignancies other than DLBCL, unless the participant had been free of the disease for ≥5 years prior to screening.
5. Participants with:

   * positive hepatitis B and/or C serology.
   * known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV)
   * CNS lymphoma involvement
   * history or evidence of clinically significant cardiovascular, CNS and/or other systemic disease that would in the investigator's opinion preclude participation in the study or compromised the participant's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Duell, MD, Principal Investigator — MorphoSys AG
Locations (57):
- United States (10):
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - UCLA - David Geffen School of Medicine, Los Angeles, California
  - Cancer Care - Torrance Memorial Physician Network, Redondo Beach, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - St. Mary's Hospital And Regional Medical Center, Grand Junction, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - St. Joseph Mercy Hospital Cancer Care Center, Ypsilanti, Michigan
  - Ohio State University Medical Center, Columbus, Ohio
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Tyler Hematology-Oncology, Tyler, Texas
- Belgium (4):
  - ZNA Middelheim dep Klinische studies Hematologie, Antwerp
  - AZ Groeninge-Campus Maria's Voorzienigheid, Kortrijk
  - Centre Hospitalier Universitaire (CHU) de Liege, Liège
  - Clinique Universitaire de Mont Godinne, Yvoir
- University Hospital Olomouc Hematoonkologicka klinika, Olomouc, Czechia
- France (4):
  - CHU De Clermont Ferrand - Hopital Estaing Service Hematologie Clinique Et Thrapie Cellulaire, Clermont-Ferrand
  - Centre Hospitalier Universitaire (CHU) De Limoges Hopital Dupuytren, Limoges
  - Centre Hospitalier Lyon-Sud (CHLS), Lyon
  - Hopital Universitaire Necker Enfants Malades Service de Hematologie Adultes, Paris
- Germany (5):
  - Universitatsklinikum Essen, Abteilung Haematologie, Essen
  - Krankenhaus Nordwest GmbH - Institut Fuer Klinisch-Onkologische Forschung (IKF), Frankfurt
  - Klinikum Grosshadern-Klinikum Der Ludwig-Maximilian Universitaet Muenchen, Munich
  - Klinikum Nuernberg Nord Medizinische Klinik 5 Hamatologie, Nuremberg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (4):
  - Semmelweis Egyetem I. Sz. Belgyogyaszati Klinika-Semmelweis University, Budapest
  - National Institute of Oncology Hematological Department, Budapest
  - DEKK, Belgyogyaszati Klinika, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz (Kaposi Mor County Hospital), Kaposvár
- Italy (9):
  - Azienda Ospedaliera Univerisitaria Policlinico Consorziale Di Bari UOC Ematologia con Trapianto, Bari
  - Ist.Ematologia E Oncologia Medica L.E A.Seragnoli Azienda Ospedaliero-Universitaria, Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Careggi-S.O.D. Patologia Medica, Florence
  - Azienda Ospedaliero - Universitaria Policlinico di Modena Dip di Medicina Diagnostica, Clinica e di Sanità Pubblica, Modena
  - AOU Maggiore della Cartia, Novara
  - A .O. S. Maria della Misericordia, Perugia
  - Tor Vergata University Department Of Hematology, Roma
  - Az Ospedaliera Santa Maria Facolta di Medicina e Chirurgia, Terni
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino
- Poland (8):
  - Pratia MCM Krakow, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSWiA z Warmimsko, Olsztyn
  - Szpital Wojewodzk I w Opolu SP ZOZ Oddzial Hematologii i Onkologii Hematologicznej, Opole
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych w Poznaniu im. prof. Ludwika Bierkowskiego, Poznan
  - Szpital Wojewodzki Nr 1 im. Fryderyka Chopina w Rzeszowie, Rzeszów
  - MTZ Clinical Research Sp. z o.o, Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy Klinika Nowotworow Ukladu Chlonnego Ul., Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol (HUGTP), Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala D'Oncologia-Hospital Duran Y Reynals, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz Servicio de Hematologia Unidad de Linformas Oncohealth Institute, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Complejo Hospitalario de Navarra (CHN), Pamplona
  - Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón
  - Hospital Universitario Virgen del Rocio, Hospital de la Mujer Servicio de Hematologia, Seville
- United Kingdom (4):
  - The Royal Bournemouth & Christchurch Hospitals, Bournemouth
  - Royal Liverpool University Hospital - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Sarah Cannon Research Institute, London
  - The Newcastle Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Salles G, Duell J, Gonzalez Barca E, Tournilhac O, Jurczak W, Liberati AM, Nagy Z, Obr A, Gaidano G, Andre M, Kalakonda N, Dreyling M, Weirather J, Dirnberger-Hertweck M, Ambarkhane S, Fingerle-Rowson G, Maddocks K. Tafasitamab plus lenalidomide in relapsed or refractory diffuse large B-cell lymphoma (L-MIND): a multicentre, prospective, single-arm, phase 2 study. Lancet Oncol. 2020 Jul;21(7):978-988. doi: 10.1016/S1470-2045(20)30225-4. Epub 2020 Jun 5. PMID 32511983
- [Result] Duell J, Maddocks KJ, Gonzalez-Barca E, Jurczak W, Liberati AM, De Vos S, Nagy Z, Obr A, Gaidano G, Abrisqueta P, Kalakonda N, Andre M, Dreyling M, Menne T, Tournilhac O, Augustin M, Rosenwald A, Dirnberger-Hertweck M, Weirather J, Ambarkhane S, Salles G. Long-term outcomes from the Phase II L-MIND study of tafasitamab (MOR208) plus lenalidomide in patients with relapsed or refractory diffuse large B-cell lymphoma. Haematologica. 2021 Sep 1;106(9):2417-2426. doi: 10.3324/haematol.2020.275958. PMID 34196165
- [Result] Duell J, Obr A, Augustin M, Endell J, Liu H, Geiger S, Silverman IM, Ambarkhane S, Rosenwald A. CD19 expression is maintained in DLBCL patients after treatment with tafasitamab plus lenalidomide in the L-MIND study. Leuk Lymphoma. 2022 Feb;63(2):468-472. doi: 10.1080/10428194.2021.1986219. Epub 2021 Nov 15. No abstract available. PMID 34779360
- [Derived] Duell J, Abrisqueta P, Andre M, Gaidano G, Gonzales-Barca E, Jurczak W, Kalakonda N, Liberati AM, Maddocks KJ, Menne T, Nagy Z, Tournilhac O, Kuffer C, Bakuli A, Amin A, Gurbanov K, Salles G. Tafasitamab for patients with relapsed or refractory diffuse large B-cell lymphoma: final 5-year efficacy and safety findings in the phase II L-MIND study. Haematologica. 2024 Feb 1;109(2):553-566. doi: 10.3324/haematol.2023.283480. PMID 37646664
- [Derived] Cherng HJ, Westin JR. Broadening the MIND: Tafasitamab and Lenalidomide versus Synthetic Controls. Clin Cancer Res. 2022 Sep 15;28(18):3908-3910. doi: 10.1158/1078-0432.CCR-22-1626. PMID 35861632
- [Derived] Nowakowski GS, Yoon DH, Peters A, Mondello P, Joffe E, Fleury I, Greil R, Ku M, Marks R, Kim K, Zinzani PL, Trotman J, Huang D, Waltl EE, Winderlich M, Kurukulasuriya NC, Ambarkhane S, Hess G, Salles G. Improved Efficacy of Tafasitamab plus Lenalidomide versus Systemic Therapies for Relapsed/Refractory DLBCL: RE-MIND2, an Observational Retrospective Matched Cohort Study. Clin Cancer Res. 2022 Sep 15;28(18):4003-4017. doi: 10.1158/1078-0432.CCR-21-3648. PMID 35674661
- [Derived] Zinzani PL, Rodgers T, Marino D, Frezzato M, Barbui AM, Castellino C, Meli E, Fowler NH, Salles G, Feinberg B, Kurukulasuriya NC, Tillmanns S, Parche S, Dey D, Fingerle-Rowson G, Ambarkhane S, Winderlich M, Nowakowski GS. RE-MIND: Comparing Tafasitamab + Lenalidomide (L-MIND) with a Real-world Lenalidomide Monotherapy Cohort in Relapsed or Refractory Diffuse Large B-cell Lymphoma. Clin Cancer Res. 2021 Nov 15;27(22):6124-6134. doi: 10.1158/1078-0432.CCR-21-1471. Epub 2021 Aug 25. PMID 34433649
- See also: CD19 expression is maintained in DLBCL patients after treatment with tafasitamab plus lenalidomide in the L-MIND study — https://pubmed.ncbi.nlm.nih.gov/34779360/
- See also: Tafasitamab plus lenalidomide in relapsed or refractory diffuse large B-cell lymphoma (L-MIND): a multicentre, prospective, single-arm, phase 2 study — https://pubmed.ncbi.nlm.nih.gov/32511983/
- See also: Long-term outcomes from the Phase II L-MIND study of tafasitamab (MOR208) plus lenalidomide in patients with relapsed or refractory diffuse large B-cell lymphoma — https://pubmed.ncbi.nlm.nih.gov/34196165/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were enrolled into this study at sites in Hungary, Belgium, Czechia, France, Poland, Italy, Germany, Spain, United Kingdom, and the United States.
Groups:
- Treatment (MOR00208, Lenalidomide): MOR00208:
  MOR00208 was administered via IV infusion at a dose of 12 mg/kg. For the first three cycles (Cycles 1 to 3) of the study each cycle consisted of a MOR00208 infusion on Day 1, Day 8, Day 15 and Day 22 of the cycle. Additionally, a loading dose was administered on Day 4 of Cycle 1. Thereafter MOR00208 was administered on a bi-weekly (every 14 days) basis with infusions on Day 1 and Day 15 of each 28-day cycle.
  LEN:
  Participants self-administered a starting dose of 25 mg oral LEN daily on Days 1-21 of each cycle, for up to 12 cycles in total. LEN dose could be modified in a de-escalating fashion or discontinued based upon clinical and laboratory findings. On days when both study drugs were given together, LEN was administered prior to MOR00208.
Period: Overall Study
Arm/Group | Treatment (MOR00208, Lenalidomide)
Started | 81
Received MOR00208 + LEN | 80
Received MOR00208 Only | 1
Completed: Participants Who Were Still on Treatment at EOS | 8
Not Completed: Participants Who Were no Longer Receiving Treatment at EOS | 73
Completed | 8
Not Completed | 73
Not completed — Adverse Event | 16
Not completed — Death | 2
Not completed — Withdrawal by Subject | 8
Not completed — Progressive disease/ Disease relapse | 42
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (MOR00208, Lenalidomide)
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 72
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 7
  Belgium | 5
  United States | 6
  Czechia | 3
  Poland | 7
  Italy | 13
  United Kingdom | 5
  France | 9
  Germany | 11
  Spain | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Objective Response Rate (ORR)
Description: ORR = complete response [CR] + partial response [PR]; Independent Radiology/Clinical Review Committee (IRC) Evaluation.
  ORR after MOR00208 and Lenalidomide combination therapy assessed by the IRC evaluation.
  ORR was defined as the number of participants of the total number of participants treated with MOR00208 + LEN with CR or PR as best response achieved at any time during the study.
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: Full analysis set (FAS): The FAS included all participant who received at least one dose of MOR00208 and at least one dose of LEN. This meant that both study drugs had to be administered at least once.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (MOR00208, Lenalidomide): MOR00208:
  MOR00208 was administered via IV infusion at a dose of 12 mg/kg. For the first three cycles (Cycles 1 to 3) of the study each cycle consisted of a MOR00208 infusion on Day 1, Day 8, Day 15 and Day 22 of the cycle.
  Additionally, a loading dose was administered on Day 4 of Cycle 1. Thereafter MOR00208 was administered on a bi-weekly (every 14 days) basis with infusions on Day 1 and Day 15 of each 28-day cycle.
  LEN:
  Participants self-administered a starting dose of 25 mg oral LEN daily on Days 1-21 of each cycle, for up to 12 cycles in total. LEN dose could be modified in a de-escalating fashion or discontinued based upon clinical and laboratory findings.
Arm/Group | Treatment (MOR00208, Lenalidomide)
Number analyzed (Participants) | 80
Participants
  Approximately 4.5 years after first participant enrolled | 46
  Approximately 6.5 years after first participant enrolled | 46

2. Secondary Outcome: Duration of Response (DoR) by IRC Evaluation
Description: DoR [months] = (date of assessment of tumor progression or death - date of assessment of first documented response of (CR or PR) + 1)/30.4375.
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: FAS: The FAS included all participants who received at least one dose of MOR00208 and at least one dose of LEN. This meant that both study drugs had to be administered at least once. Inclusive of participants with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (MOR00208, Lenalidomide)
Number analyzed (Participants) | 46
Months
  Approximately 4.5 years after first participant enrolled | 43.9 [26.1 to NA] — [Not available]. Upper limit not reached due to insufficient number of events at later stages of follow-up.
  Approximately 6.5 years after first participant enrolled | NA [33.8 to NA] — [Not available]. Median and upper limit not reached due to insufficient number of events at later stages of follow-up.

3. Secondary Outcome: DoR by Investigator (INV) Evaluation
Description: DoR [months] = (date of assessment of tumour progression or death - date of assessment of first documented response of (CR or PR) + 1)/30.4375.
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Tafasitamab (MOR00208) + Lenalidomide (LEN): MOR00208:
  MOR00208 was administered via IV infusion at a dose of 12 mg/kg. For the first three cycles (Cycles 1 to 3) of the study each cycle consisted of a MOR00208 infusion on Day 1, Day 8, Day 15 and Day 22 of the cycle.
  Additionally, a loading dose was administered on Day 4 of Cycle 1. Thereafter MOR00208 was administered on a bi-weekly (every 14 days) basis with infusions on Day 1 and Day 15 of each 28-day cycle.
  LEN:
  Participants self-administered a starting dose of 25 mg oral LEN daily on Days 1-21 of each cycle, for up to 12 cycles in total. LEN dose could be modified in a de-escalating fashion or discontinued based upon clinical and laboratory findings.
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 52
Months
  Approximately 4.5 years after first participant enrolled | 43.9 [13.9 to NA] — Not available. Upper limit not reached due to insufficient number of events at later stages of follow-up.
  Approximately 6.5 years after first participant enrolled | 43.4 [14.1 to NA] — Not available. Upper limit not reached due to insufficient number of events at later stages of follow-up.

4. Secondary Outcome: Progression-free Survival (PFS) by IRC Evaluation
Description: PFS time was defined as the time (in months) from the date of the first administration of any study drug to the date of tumor progression or death from any cause.
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 42
Months
  Approximately 4.5 years after first participant enrolled | 11.6 [6.3 to 45.7]
  Approximately 6.5 years after first participant enrolled | 11.6 [5.7 to 45.7]

5. Secondary Outcome: PFS by INV Evaluation
Description: as for outcome 4
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: FAS: The FAS includes all participants who received at least one dose of MOR00208 and one dose of LEN. This meant that both study drugs had to be administered at least once. Inclusive of participants with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 49
Months
  Approximately 4.5 years after first participant enrolled: number analyzed (Participants) | 46
  Approximately 4.5 years after first participant enrolled | 9.1 [5.5 to 28.0]
  Approximately 6.5 years after first participant enrolled | 9.1 [5.5 to 45.5]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first administration of any study drug until death from any cause (documented by the date of death).
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: FAS: The FAS includes all participants who received at least one dose of MOR00208 and one dose of LEN. This means that both study drugs must have been applied at least once. Inclusive of participants with available data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 44
Months
  Approximately 4.5 years after first participant enrolled: number analyzed (Participants) | 41
  Approximately 4.5 years after first participant enrolled | 33.5 [18.3 to NA] — Not available. Upper limit not reached due to insufficient number of events at later stages of follow-up.
  Approximately 6.5 years after first participant enrolled | 33.5 [18.3 to NA] — Not available. Upper limit not reached due to insufficient number of events at later stages of follow-up.

7. Secondary Outcome: Disease Control Rate (DCR) by IRC Evaluation
Description: DCR = CR + PR + SD (Stable disease); IRC Evaluation DCR was defined as the number of participants having CR, PR or SD based on the best objective response achieved at any time during the study.
Time Frame: Approximately 2.5 years after first participant enrolled
Population: FAS: The FAS included all participants who received at least one dose of MOR00208 and at least one dose of LEN. This meant that both study drugs had to be administered at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 80
Participants | 59

8. Secondary Outcome: DCR by INV Evaluation
Description: as for outcome 7
Time Frame: Approximately 2.5 years after first participant enrolled
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 80
Participants | 60

9. Secondary Outcome: Time to Progression (TTP) by IRC Evaluation
Description: TTP is defined as the time from the first administration of any study drug until documented DLBCL progression or death as a result of lymphoma.
Time Frame: Approximately 2.5 years after first participant enrolled
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 35
Months | 16.2 [7.4 to NA] — Not available. Upper limit not reached due to insufficient number of events at later stages of follow-up.

10. Secondary Outcome: TTP by INV Evaluation
Description: as for outcome 9
Time Frame: Approximately 2.5 years after first participant enrolled
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 40
Months | 14.1 [6.3 to NA] — Not available. Upper limit not reached due to insufficient number of events at later stages of follow-up.

11. Secondary Outcome: Time to Next Treatment (TTNT)
Description: Kaplan-Meier analysis of TTNT in FAS population. TTNT is defined as the time from the first administration of any study drug to the institution of next anti-neoplastic therapy (for any reason including disease progression, treatment toxicity and participant preference) or death of any cause, whatever comes first.
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 55
Months
  Approximately 4.5 years after first participant enrolled: number analyzed (Participants) | 51
  Approximately 4.5 years after first participant enrolled | 12.1 [7.3 to 24.7]
  Approximately 6.5 years after first participant enrolled | 12.5 [7.3 to 28]

12. Secondary Outcome: Event-free Survival (EFS) by IRC Evaluation
Description: EFS is defined as the time (in months) from the date of the first administration of any study drug to the date of tumour progression, first initiation of a new non-study anti-neoplastic therapy or death from any cause whichever comes first.
Time Frame: Approximately 4.5 years after first participant enrolled; Approximately 6.5 years after first participant enrolled
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 55
Months
  Approximately 4.5 years after first participant enrolled: number analyzed (Participants) | 53
  Approximately 4.5 years after first participant enrolled | 8.7 [5.3 to 21.0]
  Approximately 6.5 years after first participant enrolled | 9.1 [5.3 to 23.5]

13. Secondary Outcome: Serum Drug Levels of MOR00208
Description: The pharmacokinetics (PK) profile of MOR00208 was investigated by quantifying serum drug levels at baseline and after repeated IV administrations for up to 24 treatment cycles using sparse sampling.
  MOR00208 PK sample was taken pre-dose and 1 hour ± 10 min after the end of MOR00208 infusion for Cycle 1 to Cycle 23. MOR00208 PK sample (pre-dose only) were taken in odd numbered additional treatment cycles only (e.g., treatment Cycles 13, 15,17, 19, 21, 23).
Time Frame: Cycle 1 Days 1, 4, 15 predose and 1 hr post-dose; Cycle 2 Days 1, 15 predose and 1 hr post-dose; Cycle 3 Days 1, 15 predose and 1 hr post-dose; Cycles 4, 5, 6, 7, 9, 11,13, 15, 17, 19, 21, 23 Day 1 predose; End of Treatment
Population: PK analysis set (PKAS): The PKAS included all participants who received at least one dose of MOR00208 and had at least one quantifiable MOR00208 serum concentration.
  Number analyzed includes only participants with data at each timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 81
ng/mL
  Cycle 1 Day 1 (Predose): number analyzed (Participants) | 79
  Cycle 1 Day 1 (Predose) | 6.7 (53.09)
  Cycle 1 Day 1 (1 hour post dose): number analyzed (Participants) | 71
  Cycle 1 Day 1 (1 hour post dose) | 249075.9 (53724.93)
  Cycle 1 Day 4 (pre-dose): number analyzed (Participants) | 73
  Cycle 1 Day 4 (pre-dose) | 126306.8 (39105.37)
  Cycle 1 Day 4 (1 hour post-dose): number analyzed (Participants) | 65
  Cycle 1 Day 4 (1 hour post-dose) | 363626.2 (82971.54)
  Cycle 1 Day 15 (pre dose): number analyzed (Participants) | 75
  Cycle 1 Day 15 (pre dose) | 157722.3 (50655.86)
  Cycle 1 Day 15 (1 hour post-dose): number analyzed (Participants) | 70
  Cycle 1 Day 15 (1 hour post-dose) | 396262.1 (97215.09)
  Cycle 2 Day 1 (predose): number analyzed (Participants) | 71
  Cycle 2 Day 1 (predose) | 181870.8 (72582.62)
  Cycle 2 Day 1 (1 hour post-dose): number analyzed (Participants) | 62
  Cycle 2 Day 1 (1 hour post-dose) | 439788.2 (126930.55)
  Cycle 2 Day 15 (Pre Dose): number analyzed (Participants) | 63
  Cycle 2 Day 15 (Pre Dose) | 217846.9 (77799.93)
  Cycle 2 Day 15 (1 hour post-dose) ): number analyzed (Participants) | 59
  Cycle 2 Day 15 (1 hour post-dose) ) | 442940.2 (85475.90)
  Cycle 3 Day 1 (predose): number analyzed (Participants) | 61
  Cycle 3 Day 1 (predose) | 208520.6 (68866.46)
  Cycle 3 Day 1 (1 hour post-dose): number analyzed (Participants) | 53
  Cycle 3 Day 1 (1 hour post-dose) | 466135.8 (112647.31)
  Cycle 3 Day 15 (predose): number analyzed (Participants) | 51
  Cycle 3 Day 15 (predose) | 223909.4 (85170.91)
  Cycle 3 Day 15 (1 hour post-dose): number analyzed (Participants) | 44
  Cycle 3 Day 15 (1 hour post-dose) | 455635.0 (104198.64)
  Cycle 4 Day 1 (predose) ): number analyzed (Participants) | 52
  Cycle 4 Day 1 (predose) ) | 216328.4 (94553.25)
  Cycle 5 Day 1 (pre dose): number analyzed (Participants) | 51
  Cycle 5 Day 1 (pre dose) | 142134.4 (72691.16)
  Cycle 6 Day 1 (pre dose): number analyzed (Participants) | 49
  Cycle 6 Day 1 (pre dose) | 115132.3 (55774.77)
  Cycle 7 Day 1 (pre dose): number analyzed (Participants) | 49
  Cycle 7 Day 1 (pre dose) | 114661.5 (73328.15)
  Cycle 9 Day 1 (pre dose): number analyzed (Participants) | 40
  Cycle 9 Day 1 (pre dose) | 108640.4 (52282.72)
  Cycle 11 Day 1 (pre dose): number analyzed (Participants) | 34
  Cycle 11 Day 1 (pre dose) | 126472.0 (64872.47)
  Cycle 13 Day 1 (pre dose): number analyzed (Participants) | 31
  Cycle 13 Day 1 (pre dose) | 100853.5 (61229.42)
  Cycle 15 Day 1 (pre dose): number analyzed (Participants) | 30
  Cycle 15 Day 1 (pre dose) | 159676.5 (61199.32)
  Cycle 17 Day 1 (pre dose): number analyzed (Participants) | 25
  Cycle 17 Day 1 (pre dose) | 175855.1 (64592.17)
  Cycle 19 Day 1 (pre dose): number analyzed (Participants) | 21
  Cycle 19 Day 1 (pre dose) | 197045.0 (69962.05)
  Cycle 21 Day 1 (pre dose): number analyzed (Participants) | 19
  Cycle 21 Day 1 (pre dose) | 197228.0 (53222.03)
  Cycle 23 Day 1 (pre dose): number analyzed (Participants) | 15
  Cycle 23 Day 1 (pre dose) | 224253.3 (64686.85)
  End of Treatment: number analyzed (Participants) | 39
  End of Treatment | 141240.7 (114804.40)

14. Secondary Outcome: Number of Participants Who Developed Anti-MOR00208 Antibodies
Description: The Anti-MOR00208 Antibodies were investigated by quantifying serum drug levels at baseline and after repeated intravenous (IV) administrations planned for up to 24 treatment cycles using sparse sampling. Anti-MOR00208 antibody sample (pre-dose only) were taken in odd numbered additional treatment cycles only (e.g., treatment Cycles 13, 15,17, 19, 21,23).
Time Frame: Baseline, Up to a maximum of 23 cycles.
Population: Immunogenicity analysis set (IAS): The IAS included participants who had at least one anti-MOR00208 antibody assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 81
Participants
  Yes (Treatment-emergent ADAs) | 0
  No (Negative baseline and post baseline results) | 72
  Not evaluable (Positive baseline results) | 2
  Missing (No post baseline results available) | 7

15. Secondary Outcome: Number of Participants That Experienced Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are defined as any adverse event reported in the following time interval (including the lower and upper limits): date of first administration of study treatment; date of last administration of study treatment + 30 days, or if they are considered to be related to the study drug.
Time Frame: Approximately 6.5 years after first participant enrolled
Population: Safety analysis set (SAF):
  The SAF includes all participants who received at least one dose of MOR00208 or LEN and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 81
Participants | 81

16. Secondary Outcome: Severity of Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with Severity of TEAEs during MOR00208 and LEN combination therapy.
Time Frame: Approximately 6.5 years after first participant enrolled
Population: SAF:
  The SAF includes all participants who received at least one dose of MOR00208 or LEN and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tafasitamab (MOR00208) + Lenalidomide (LEN)
Number analyzed (Participants) | 81
Participants
  Severe | 43
  Moderate | 31
  Mild | 6
  Missing | 1

ADVERSE EVENTS:
Time Frame: From first day of study drug administration through 30 days after last dose, up to maximum duration of 6.5 years approximately after first participant enrolled.
Description: All adverse events (AEs) (except non-serious AEs for screening failures) that occurred after the provision of informed consent and up to 30 days after last study drug administration was recorded in the eCRF and in the participant's medical records, whether or not they were considered by the investigator to be related to the study drug. Thereafter, only AEs assessed as related were collected at the end of the study.
Groups:
- Treatment (MOR00208, Lenalidomide): MOR00208 was administered via intravenous Infusion, weekly (Cycle 1-3) of the study each cycle consisted of a MOR00208 infusion on Day 1, Day 8, Day 15 and Day 22 of the cycle. Additionally, a loading dose was administered on Day 4 of Cycle 1. Thereafter MOR00208 was administered on a bi-weekly (every 14 days) basis with infusions on Day 1 and Day 15 of each 28-day cycle, until disease progression or unacceptable toxicity or discontinuation due to any other reason.
  Lenalidomide (Revlimid®), PO, daily, on Days 1-21 of each cycle, for up to 12 cycles in total. LEN dose could be modified in a de-escalating fashion or discontinued based upon clinical and laboratory findings. Treatment with LEN was stopped in case of disease progression, or unacceptable toxicity, or discontinuation for any other reason.
  On days when both study drugs were given together, LEN was administered prior to tafasitamab.
Arm/Group | Treatment (MOR00208, Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 45/81
Serious Adverse Events (participants affected / at risk) | 47/81
Other Adverse Events (participants affected / at risk) | 75/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (MOR00208, Lenalidomide) (N=81)
Pneumonia (Infections and infestations) | 7 (7)
Bronchitis (Infections and infestations) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (4)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2)
Haematoma (Vascular disorders) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (MOR00208, Lenalidomide) (N=81)
Neutropenia (Blood and lymphatic system disorders) | 40 (215)
Anaemia (Blood and lymphatic system disorders) | 30 (74)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (71)
Leukopenia (Blood and lymphatic system disorders) | 10 (44)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6)
Lymphopenia (Blood and lymphatic system disorders) | 5 (10)
Diarrhoea (Gastrointestinal disorders) | 30 (63)
Constipation (Gastrointestinal disorders) | 15 (21)
Nausea (Gastrointestinal disorders) | 12 (21)
Vomiting (Gastrointestinal disorders) | 12 (15)
Abdominal pain (Gastrointestinal disorders) | 8 (9)
Asthenia (General disorders) | 21 (39)
Oedema peripheral (General disorders) | 20 (35)
Pyrexia (General disorders) | 18 (39)
Fatigue (General disorders) | 13 (24)
Mucosal inflammation (General disorders) | 6 (9)
Bronchitis (Infections and infestations) | 12 (19)
Nasopharyngitis (Infections and infestations) | 8 (11)
Respiratory tract infection (Infections and infestations) | 9 (17)
Upper respiratory tract infection (Infections and infestations) | 8 (9)
Urinary tract infection (Infections and infestations) | 10 (15)
Gastroenteritis (Infections and infestations) | 6 (9)
Decreased appetite (Metabolism and nutrition disorders) | 18 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 15 (28)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (26)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (19)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (913)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
C-reactive protein increased (Investigations) | 9 (12)
Blood creatinine increased (Investigations) | 7 (17)
Gamma-glutamyltransferase increased (Investigations) | 6 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 8 (10)
Headache (Nervous system disorders) | 7 (19)
Paraesthesia (Nervous system disorders) | 7 (7)
Hypertension (Vascular disorders) | 7 (10)
Hypotension (Vascular disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 6 (10)
Hypogammaglobulinaemia (Immune system disorders) | 5 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (5)
Dysuria (Renal and urinary disorders) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 5 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Sciatica (Nervous system disorders) | 5 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (18)
Rhinitis (Infections and infestations) | 7 (7)
Sinusitis (Infections and infestations) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT02399085/Prot_001.pdf
  • Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT02399085/SAP_002.pdf